CLINICAL TRIAL: NCT04160962
Title: A Real World Study of the Effect of Laparoscopic Preservation of the Pylorus and Vagus Nerve on the Postoperative Quality of Life in Patients With Early Gastric Cancer
Brief Title: A Real World Study of Laparoscopic Preservation of the Pylorus Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LAPPG RWS
Record Dates: First submitted 2019-11-04; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lappg
  Interventions: Procedure: lappg
- ladgbi
  Interventions: Procedure: lappg

INTERVENTIONS:
Procedure: lappg — Laparoscopic gastrectomy for pylorus preservation

SUMMARY:
For the patients with early gastric cancer (T1), preoperative evaluation (gastroscope, ultrasound gastroscope and abdominal enhanced CT) showed that the tumor was located in the body of the stomach, and the margin was enough to retain the pylorus and non lymph node metastasis (N0). Lappg (D1 + lymph node dissection) and traditional laparoscopic distal gastrectomy (BII type anastomosis, D1 + lymph node dissection) were included A control study was conducted to evaluate the difference of long-term quality of life, gastric emptying rate, incidence of basic reflux gastritis, bile contraction function, immune index, nutritional index and disease-free survival and overall survival between the two groups.

DETAILED DESCRIPTION:
The overall design of this study is an experimental study based on the real world. All the patients in the study group were from early gastric cancer patients who were operated on in gastrointestinal surgery of Renji Hospital. According to the preoperative evaluation of early gastric cancer (gastroscope, ultrasonic gastroscope and abdominal enhanced CT), patients with early gastric cancer whose tumor is located in the gastric body and whose cutting edge is enough to retain pylorus and non lymph node metastasis (N0) were included in the study. Group A (Study Group): lappg treatment group, group B (control group): laparoscopic distal gastrectomy type I group. In this study, group A was taken as the study group and group B as the control group Group, the differences between groups were compared. The main end point was the quality of life score (eortc-qlq-c30 scale, see the attached table). According to the literature and the data of the retrospective study of the center, it was assumed that the expected mean of the study group after treatment was 7.27, the mean of the control group after treatment was 6.76, and the total standard deviation of the test group and the control group was 0.51. The design of the test group and the control group was 1:1. According to this, two independent α = 0.05 were carried out Test of the average number of standing samples. It is calculated that 144 patients (72 in each group) are needed, so that under the test level of α = 0.05, according to 80% test efficiency, the difference between the two groups is statistically significant. Assuming that 10% of the patients could not be evaluated (shedding), 80 patients in each group were enrolled, and 160 patients in both groups were enrolled.

2) inclusion / exclusion / withdrawal criteria of subjects

Inclusion criteria: 18 years old < age < 75 years old; primary gastric lesions were diagnosed as gastric adenocarcinoma by tissue biopsy; preoperative clinical stage was T1N0M0 according to ajcc-7thtnm tumor stage; the tumor site was expected to receive R0 after pylorus preserving gastrectomy and D1 + lymph node dissection; preoperative Eastern Cooperative Oncology Group physical state score was 0 / 1; preoperative ASA score was I-III, with informed consent of the patient.

Exclusion criteria: pregnant or lactating women; severe mental illness; history of upper abdominal surgery (except for laparoscopic cholecystectomy); history of gastric surgery (including endoscopic submucosal dissection/ endoscopic mucosal resection for gastric cancer); preoperative imaging examination showed regional enlarged lymph nodes; history of other malignant diseases within 5 years; patients with gastric cancer who have implemented new adjuvant treatment or recommended new adjuvant treatment; no History of stable angina pectoris or myocardial infarction; history of cerebral infarction or cerebral hemorrhage within 6 months; history of continuous systemic corticosteroid therapy within 1 month; simultaneous operation for other diseases; emergency operation for gastric cancer with complications (hemorrhage, perforation, obstruction).

Withdrawal criteria: conversion to laparotomy; intraoperative / postoperative pathological confirmation of tumor invasion depth exceeding T1, or tumor invasion of duodenum; intraoperative / postoperative pathological confirmation of lymph node metastasis; intraoperative / postoperative pathological confirmation of M1 cases; intraoperative confirmation of failure to complete D1 + lymph node dissection / R0 due to tumor reasons; intraoperative confirmation of the need for total gastrectomy to ensure safe proximity; need for other diseases During the same period of the study, the patients were operated at the same time; because of severe complications (unable to tolerate surgery or anesthesia) during the perioperative period, the treatment plan of the study was not suitable or could not be implemented according to the plan; after entering the study, because of the patient's condition change, the emergency operation was confirmed by the doctor in charge; at any stage after entering the study, the patients voluntarily requested to withdraw or suspend the treatment due to the patient's personal reasons Treatment; treatment proven to be in violation of this protocol.

3) end point of study

Primary endpoint: 5-year quality of life assessment [time window: 5 years after operation]. Secondary endpoint: 3-year quality of life [time window: 3 years after operation]; immune index [time window: 5 years after operation]; nutritional index [time window: 5 years after operation]; gastric emptying rate [time window: 5 years after operation]; incidence of basic reflux gastritis [time window: 5 years after operation]; gallbladder contraction function [time window: 5 years after operation]; 5-year total survival rate [time window: 5 years after operation] 5 years; 5-year recurrence free survival [time window: 5 years after operation].

4) diagnostic criteria for this study

In this study, ajcc-7th primary tumor, regional nodes, metastasis tumor staging system was used; the diagnostic criteria and classification of gastric cancer were based on the international diagnostic criteria of histopathology; the definition of early gastric cancer: tumor infiltration was limited to the mucosa and submucosa, and did not invade the muscular layer (T1); in this study, T1N0 was the study object, but not the study object.

5) interventions

According to the preoperative evaluation (gastroscope, ultrasonic gastroscope and abdominal enhanced CT), the tumor is located in the body of the stomach, and the cutting edge is enough to retain the pylorus and early gastric cancer without lymph node metastasis (N0). By randomized grouping, the laparoscopic pylorus preserving gastrectomy (lappg, D1 + lymphadenectomy) and traditional laparoscopic distal gastrectomy (BII type anastomosis, D1 + lymphadenectomy) are performed Bed operation intervention.

6) statistical analysis

In demographic indicators, numerical variables are mainly described by means of means and standard deviations, and classified variables are mainly described by rates or ratios. T-test, chi square test or nonparametric test can be used to test the equilibrium of two groups of demography.

Statistical analysis method of main index and secondary index. The main index is patients' postoperative quality of life score (postscript symptom scores), which is a numerical variable. The statistical description mainly uses mean and standard deviation. Statistical inference uses t-test, ANOVA or nonparametric test according to data distribution conditions. The secondary indicators involve the expression of usage rate of classified statistical description, and the expression of chi square test of statistical inference hypothesis test. If there is no balance between the two groups, we can use multiple regression to adjust the confounding factors and compare the difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1) 18 years old < age < 75 years old;

(2) primary gastric lesions were diagnosed as gastric adenocarcinoma by biopsy;

(3) the preoperative clinical stage was T1N0M0 according to ajcc-7thtnm;

(4) it is predicted that R0 can be obtained by pylorogastric gastrectomy and D1 + lymph node dissection;

(5) preoperative ECoG physical state score 0 / 1;

(6) preoperative ASA score I-III;

(7) informed consent of patients.

Exclusion Criteria:

1. pregnant or lactating women; suffering from serious mental illness;
2. the history of upper abdominal surgery (except laparoscopic cholecystectomy);
3. history of gastric surgery (including ESD / EMR for gastric cancer);
4. preoperative imaging examination showed regional enlarged lymph nodes;
5. having other malignant diseases within 5 years;
6. patients with gastric cancer who have received new adjuvant therapy or recommended new adjuvant therapy;
7. there was a history of unstable angina or myocardial infarction within 6 months;
8. have a history of cerebral infarction or cerebral hemorrhage within 6 months;
9. there was a history of continuous systemic corticosteroid therapy within 1 month;
10. simultaneous surgical treatment of other diseases is needed;
11. gastric cancer with complications (hemorrhage, perforation, obstruction) requires emergency surgery;
12. FEV1 of pulmonary function examination was less than 50% of the predicted value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the patients with early gastric cancer (T1), preoperative evaluation (gastroscope, ultrasound gastroscope and abdominal enhanced CT) showed that the tumor was located in the body of the stomach, and the margin was enough to retain the pylorus and non lymph node metastasis (N0). Lappg (D1 + lymph node dissection) and traditional laparoscopic distal gastrectomy (BII type anastomosis, D1 + lymph node dissection) were included A control study was conducted to evaluate the influence of two surgical methods on the long-term quality of life of patients after operation
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
EORTC Questionnaire QLQ-C30 | 5 years
  Among the multiple tools to evaluate QOL of postgastrectomy patients, the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30 have been used most extensively.